CLINICAL TRIAL: NCT07172646
Title: A Phase I/II, Randomized, Double Blind, Placebo Controlled, Dose-Escalation and -Expansion Study to Evaluate the Safety, Tolerability, PK, and PD of Subcutaneously Administered SRSD216 in Patients With Elevated Lipoprotein(a)
Brief Title: A Study of SRSD216 in Patients With Elevated Lipoprotein (a)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sirius Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SRSD216-101
Record Dates: First submitted 2025-08-21; First posted 2025-09-15 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Hyperlipoproteinemia (a)
MeSH Terms: conditions — Hyperlipoproteinemias

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SRSD216 injection (Part 1) (Experimental): SRSD216 administered SC. in subjects of Part 1
  Interventions: Drug: SRSD216 injection
- SRSD216 injection (Part 2) (Experimental): SRSD216 administered SC. in subjects of Part 2
  Interventions: Drug: SRSD216 injection; Drug: Placebo
- 0.9% Sodium Chloride (Part 1) (Experimental): Placbo administered SC. in subjects of Part 1
  Interventions: Drug: Placebo
- 0.9% Sodium Chloride (Part 2) (Placebo Comparator): Placbo administered SC. in subjects of Part 2
  Interventions: Drug: SRSD216 injection; Drug: Placebo

INTERVENTIONS:
Drug: SRSD216 injection — Administered SC.
  Arms: 0.9% Sodium Chloride (Part 2); SRSD216 injection (Part 1); SRSD216 injection (Part 2)
Drug: Placebo — Administered SC.
  Arms: 0.9% Sodium Chloride (Part 1); 0.9% Sodium Chloride (Part 2); SRSD216 injection (Part 2)

SUMMARY:
This is a two-part study, intended to investigate the safety, tolerability, characteristics of PK and PD of single SC dose of SRSD216 and to identify a dose range for further studies in subjects with elevated Lp(a) level with or without ASCVD history.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions;
* Males or females, of any race;
* Body mass index (BMI) between 18.0 and 40.0 kg/m2, inclusive;
* Male subjects are not allowed to donate sperm, and female subjects are not allowed to donate eggs from the time the ICF is signed until at least 3 months after the last follow-up.

Exclusion Criteria:

* Any history or evidence of abnormal bleeding or coagulopathy; or evidence of prolonged or unexplained, clinically significant bleeding, or frequent unexplained bruising or thrombosis; or history of spontaneous bleeding;
* Evidence of active or suspected cancer within 3 years prior to screening (non-melanoma skin cancer, localized prostate cancer treated with curative intent, or other in situ carcinoma that does not require systemic therapy and is considered cured for at least 1 years is allowed);
* Acute febrile illness within 7 days prior to dose administration or evidence of active infection;
* Any major surgery within 3 months prior to screening or plan to have any major surgery during the study;
* History of clinically significant hypersensitivity, intolerance, or allergy to any oligonucleotide or GalNAc as determined by the investigator;
* Fasting TG≥ 500 mg/dL (5.6 mmol/L) during screening;
* Receipt of an investigational drug within 30 days or 5 half-lives of that drug, whichever is longer, prior to dose administration in this study;
* Have previously completed or withdrawn from this study or any other study investigating SRSD216 and have previously received SRSD216.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | 1 year
  A summary of TEAE to evaluate the safety and tolerability of SRSD216

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sirius Therapeutics
Locations (1):
- Site 01, Beijing, Beijing Municipality, China